CLINICAL TRIAL: NCT01326143
Title: ORM Narval Mandibular Repositioning Device in the Second-line Treatment of Severe OSAH
Brief Title: Narval CC Mandibular Repositioning Device in the Second-line Treatment of Severe Obstructive Sleep Apnea Hypopnea (OSAH)
Acronym: ORCADES
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: RESMED Narval ORM 001; 2010-A01121-38 (Registry Identifier: ID RCB AFSSAPS)
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: MRD; Narval; Oral appliance; Obstructive Sleep apnea; OSAH; OSA treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ORM Narval MRD
  Interventions: Device: ORM Narval MRD

INTERVENTIONS:
Device: ORM Narval MRD

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy, tolerance and compliance of ORM Narval Mandibular Repositioning Device (MRD) as a second-line treatment for patients with severe Obstructive Sleep Apnea Hypopnea (OSAH) syndrome who refuse or are intolerant to Continuous Positive Airway Pressure (CPAP) treatment.

DETAILED DESCRIPTION:
OSAH is a common condition which occurs in between 1 and 4% of the adult population. Respiratory obstruction may be complete (apnea) or incomplete (hypopnea). This disorder disturbs the architecture and quality of sleep, and is a known risk factor in the development of cardiovascular and metabolic diseases. CPAP is the standard treatment, however in some cases patients are unable to use it (rejection, intolerance, etc.). In such circumstances, treatment using a MRD may result in an improvement of symptoms.

Very few long-term clinical data are available on treatment of OSAH by MRD. This study should allow to have a precise and representative vision of 5 years results of ORM Narval MRD treatment in conditions of good practices (titration, controls of efficacy).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with severe OSAH (AHI > 30 or AHI of between 5 and 30 along with severe daytime sleepiness),
* intolerant to or having refused CPAP therapy,
* no dental, parodontal or articulatory contraindications,
* no experience of any mandibular advancement device therapy,
* medical insurance.

Exclusion Criteria:

* severe psychiatric disorders or severe neuromuscular disorders
* > 20% of central apneas during the baseline assessment,
* severe OSAH with an AHI > 30 associated with another sleep pathology (narcolepsy with or without cataplexy, idiopathic hypersomnia, severe restless legs syndrome),
* pregnant or breastfeeding woman,
* Informed consent not signed,
* patient requiring special protection such as patients with appointed guardians and patients without legal or administrative rights,
* patient who is completely or partially edentulous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe Obstructive Sleep Apnea Hypopnea
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Apnea/Hypopnea Index (AHI) reduced by at least 50% compared to baseline measured by Polygraphy/Polysomnography (PG/PSG) | 5 years

SECONDARY OUTCOMES:
Percentage of patients with AHI reduced by at least 50% compared to baseline measured by PG/PSG | 3 months and 2 years
Percentage of patients who no longer suffer from severe daytime sleepiness (Epworth Sleepiness scale) | 3 months, 2 years and 5 years
Sleep quality of life (Quebec Sleep Questionaire) | 3 months, 2 years and 5 years
Percentage of patients who stopped the therapy for dento-maxillofacial side effects | 6 months, 1, 2, 3, 4 and 5 years
Percentage of patients with satisfactory compliance | 3 months, 2 and 5 years.
Fatigue score (Pichot questionaire) | 3 months, 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Françoise VECCHIERINI-BLINEAU, Dr, Principal Investigator — Hôtel Dieu, Paris
Locations (26):
- France (26):
  - Fondation Bon Sauveur / cabinet médical / cabinet dentaire, Albi
  - CH Antibes / cabinet dentaire, Antibes
  - CH Béziers, Béziers
  - CHU Avicennes, Bobigny
  - Polyclinique du Tondu / cabinet dentaire, Bordeaux
  - CHG Chalon en Champagne, Châlons-en-Champagne
  - CH Compiègne Senlis / cabinets dentaires, Compiègne
  - CHU Grenoble, Grenoble
  - Cabinet médical / cabinet dentaire, Lagny
  - CHRU Lille, Lille
  - Cabinet médical Lyon, Lyon
  - CHU La Timone / cabinet médical, Marseille
  - CHRU Montpellier / Clinique Beau Soleil / Faculté d'Odontologie / cabinet dentaire, Montpellier
  - CH Montreuil, Montreuil
  - Centre Médical Plateau de Haye / cabinet médical / cabinet dentaire, Nancy
  - Maison de la Mutualité / polyclinique de l'Atlantique, Nantes
  - Cabinet médical / cabinet dentaire, Nice
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital Pitié Salpetriere, Paris
  - Hôtel Dieu, Paris
  - CHU Poitiers, Poitiers
  - CHRU Rennes / polyclinique St Laurent / cabinet dentaire, Rennes
  - CHRU Rouen, Rouen
  - CHU Toulouse, Toulouse
  - Clinique de l'Union, Toulouse
  - CH Valence, Valence

REFERENCES:
- [Result] Vecchierini MF, Attali V, Collet JM, d'Ortho MP, El Chater P, Kerbrat JB, Leger D, Monaca C, Monteyrol PJ, Morin L, Mullens E, Pigearias B, Meurice JC; ORCADES investigators. A custom-made mandibular repositioning device for obstructive sleep apnoea-hypopnoea syndrome: the ORCADES study. Sleep Med. 2016 Mar;19:131-40. doi: 10.1016/j.sleep.2015.05.020. Epub 2015 Jun 29. PMID 26364869
- [Result] Attali V, Vecchierini MF, Collet JM, d'Ortho MP, Goutorbe F, Kerbrat JB, Leger D, Lavergne F, Monaca C, Monteyrol PJ, Morin L, Mullens E, Pigearias B, Martin F, Tordjman F, Khemliche H, Lerousseau L, Meurice JC; ORCADES investigators. Efficacy and tolerability of a custom-made Narval mandibular repositioning device for the treatment of obstructive sleep apnea: ORCADES study 2-year follow-up data. Sleep Med. 2019 Nov;63:64-74. doi: 10.1016/j.sleep.2019.04.021. Epub 2019 Jun 12. PMID 31606651
- [Derived] Vecchierini MF, Attali V, Collet JM, d'Ortho MP, Goutorbe F, Kerbrat JB, Leger D, Lavergne F, Monaca C, Monteyrol PJ, Morin L, Mullens E, Pigearias B, Martin F, Khemliche H, Lerousseau L, Meurice JC; ORCADES investigators; Abedipour D, Allard-Redon A, Aranda A, Attali V, Bavozet F, Becu M, Beruben W, Bessard J, Bonafe I, Boukhana M, Chabrol B, Chatte G, Lebret C, Collet JM, Coste O, Dumont N, Durand-Amat S, D'ortho MP, Elbaum JM, De Santerre OG, Goutorbes F, Grandjean T, Guyot W, Hammer D, Havasi C, Huet P, Kerbrat JB, Khemliche H, Koltes C, Leger D, Lacassagne L, Laur X, Lerousseau L, Liard O, Loisel C, Longuet M, Mallart A, Martin F, Merle Beral F, Meurice JC, Mokhtari Z, Monaca C, Monteyrol PJ, Muir JF, Mullens E, Muller D, Paoli C, Petit FX, Pigearias B, Pradines M, Prigent A, Putterman G, Rey M, Samama M, Tamisier R, Tiberge M, Tison C, Tordjman F, Triolet B, Vacher C, Vecchierini MF, Verain A. Sex differences in mandibular repositioning device therapy effectiveness in patients with obstructive sleep apnea syndrome. Sleep Breath. 2019 Sep;23(3):837-848. doi: 10.1007/s11325-018-1766-8. Epub 2018 Dec 22. PMID 30580418